CLINICAL TRIAL: NCT01678066
Title: A Prospective Study to Bilaterally Compare a New FDA-Approved Non-Invasive Cardiac Output Monitor in Children Undergoing General Anesthesia
Brief Title: A Prospective Study to Bilaterally Compare a Non-Invasive Cardiac Output Monitor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas Anthony Anderson, Assistant in Anesthesia, Massachusetts General Hospital
Other Study IDs: 2012P001561
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Anesthesiology; Pediatrics; General Surgery; Orthopedics; General Anesthesia; Cardiac Output
Keywords: Noninvasive cardiac output.; Pediatrics.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bilateral cardiac output: This is a prospective, non-randomized study to collect data from two noninvasive FDA-approved cardiac output monitors simultaneously in pediatric patients under general anesthesia in the operating room from age 1 month old to 8 years old with all types of medical conditions. We will enroll 50 male and female pediatric patients who are having lower abdominal and lower extremity surgery in this study so that the additional 8 EKG leads placed on the patients do not interfere with the surgical site or patient positioning.
  Interventions: Device: Bilateral cardiac output

INTERVENTIONS:
Device: Bilateral cardiac output
  Other Names: Cardiotronic ICON non-invasive cardiac output monitor

SUMMARY:
Study hypothesis: The Cardiotronic ICON non-invasive cardiac output monitor gives accurate information when placed on a patient's Right or Left side.

Summary: To simultaneously compare physiologic data collected from two non-invasive cardiac output monitors placed bilaterally on pediatric patients undergoing general anesthesia. The FDA approved Cardiotronic ICON non-invasive cardiac output monitor has been validated by the manufacturer in pediatric and adult patients with leads placed on the left side. However, sometimes the surgical site and/or patient position precludes placement of the monitor leads on the left side. In such situations it would be useful to know whether placement of the monitor's leads on a patient's right side gives accurate cardiac output data. We will prospectively collect, and compare, simultaneous physiologic data for all enrolled children using two monitors, one on the patient's right side and one on the patient's left side.

DETAILED DESCRIPTION:
Traditionally cardiac output has been estimated with thermodilution, Fick oxygen consumption or with echocardiography. Other non-invasive techniques such as analysis of arterial wave forms and measurement of expired carbon dioxide have been attempted but with variable success. Recently a new device (Cardiotronic® EC™) has been approved by the FDA for use in children of all ages including neonates. Electrical cardiometry is a new method which can continuously estimate stroke volume and left ventricular outflow to calculate cardiac output, calculate cardiac index, as well as a variety of other parameters through quantitation of changes in impedance associated with changes in the orientation of red blood cells. During diastole red cells are organized chaotically but during systole they assume a position parallel to the direction of blood flow. Thus thoracic electrical bioimpedance relate to changes in thoracic aortic blood flow and through the use of refined algorithms non-invasive measurement of cardiac output is achieved.

The height (cm), gender, weight (kg) and age of the patient are entered into the hand-held device. Eight electrodes are applied to the neck and chest at specified locations, four per device. The device records the heart rate and averages cardiac output every 10-60 heartbeats again depending upon how the device is configured.

This is a prospective, non-randomized study to collect data from two noninvasive FDA-approved cardiac output monitors simultaneously in pediatric patients under general anesthesia in the operating room from age 1 month old to 8 years old with all types of medical conditions. We will enroll 50 male and female pediatric patients who are having lower abdominal and lower extremity surgery in this study so that the additional 8 EKG leads placed on the patients do not interfere with the surgical site or patient positioning.

ELIGIBILITY:
Inclusion Criteria:

* 1 month old to 8 years old.
* Lower abdominal or lower extremity surgery.

Exclusion Criteria:

* Less than 1 month old.
* Greater than 8 years old.
* Patients undergoing upper abdominal, thoracic, upper extremity, or head/neck surgery.

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who will undergo general anesthesia in the operating room from age 1 month old to 8 years old with all types of medical conditions who are having lower abdominal and lower extremity surgery in this study so that the additional 8 EKG leads placed on the patients do not interfere with the surgical site or patient positioning.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Bilateral cardiac output using the Cardiotronic ICON non-invasive cardiac output monitor. | 6 months
  To simultaneously compare physiologic data collected from two non-invasive cardiac output monitors placed bilaterally on pediatric patients undergoing general anesthesia. The FDA approved Cardiotronic ICON non-invasive cardiac output monitor has been validated by the manufacturer in pediatric and adult patients with leads placed on the left side. However, sometimes the surgical site and/or patient position precludes placement of the monitor leads on the left side. In such situations it would be useful to know whether placement of the monitor's leads on a patient's right side gives accurate cardiac output data. We will prospectively collect, and compare, simultaneous physiologic data for all enrolled children using two monitors, one on the patient's right side and one on the patient's left side.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Anderson, PhD, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Suttner S, Schollhorn T, Boldt J, Mayer J, Rohm KD, Lang K, Piper SN. Noninvasive assessment of cardiac output using thoracic electrical bioimpedance in hemodynamically stable and unstable patients after cardiac surgery: a comparison with pulmonary artery thermodilution. Intensive Care Med. 2006 Dec;32(12):2053-8. doi: 10.1007/s00134-006-0409-x. Epub 2006 Oct 13. PMID 17039348 (Retraction: PMID 21604011 Intensive Care Med. 2011 Jul;37(7):1232)
- [Background] Norozi K, Beck C, Osthaus WA, Wille I, Wessel A, Bertram H. Electrical velocimetry for measuring cardiac output in children with congenital heart disease. Br J Anaesth. 2008 Jan;100(1):88-94. doi: 10.1093/bja/aem320. Epub 2007 Nov 16. PMID 18024954
- [Background] Zoremba N, Bickenbach J, Krauss B, Rossaint R, Kuhlen R, Schalte G. Comparison of electrical velocimetry and thermodilution techniques for the measurement of cardiac output. Acta Anaesthesiol Scand. 2007 Nov;51(10):1314-9. doi: 10.1111/j.1399-6576.2007.01445.x. PMID 17944633